CLINICAL TRIAL: NCT04278911
Title: Effect of Cognitive Impairment (CI) on Prognosis in the Elderly Patients With Acute Coronary Syndrome (ACS)
Brief Title: Effect of CI on Prognosis in the Elderly Patients With ACS
Acronym: CIACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hongwei Li, MD, Prof., Beijing Friendship Hospital
Other Study IDs: BFH--CI and ACS
Record Dates: First submitted 2020-02-19; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Acute Coronary Syndrome; Cognitive Impairment; Elderly
MeSH Terms: conditions — Acute Coronary Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participates: This is an observational study
  Interventions: Diagnostic Test: MMSE and MoCA

INTERVENTIONS:
Diagnostic Test: MMSE and MoCA — This is an observational study. All the patients evaluate with MMSE (Mini-mental State Examination) and MoCA (Montreal Cognitive Assessment), and investigate the incidence and characteristics of cognitive and MACE

SUMMARY:
This study aims to investigate the incidence and characteristics of cognitive Impairment(CI) in the elderly patients with acute coronary syndrome (ACS), and to determine whether CI are predictive of the prognosis of major adverse cardiovascular events (MACE) and mortality.

ELIGIBILITY:
Inclusion Criteria:

* ≥65yr
* Confirmed ACS diagnosis （include unstable angina, ST-segment elevation myocardial infarction and Non ST-segment elevation myocardial infarction）
* fulfilled MMSE or MoCA
* patients agreed and provided informed consent

Exclusion Criteria:

* Type 2 myocardial infarction and Acute nonischemic myocardial injury
* past history of malignant tumors
* Past history of stroke or dementia
* Hepatic insufficiency (ALT>8ULN or ALT>3ULN and TBIL>2ULN)
* Renal insufficiency (GFR<15 ml/min/1.73m2)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients (≥65yr) admitted to Beijing Friendship Hospital,Capital Medical University with a confirmed ACS diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
MACE (major adverse cardiovascular events) | 12 months
  Myocardial infarction, revascularization, stroke, cardiac death, all cause of death

SECONDARY OUTCOMES:
Cognitive level decline | 12 months
  Evaluate with MMSE (Mini-mental State Examination)
Cognitive level decline | 12 months
  Evaluate MoCA (Montreal Cognitive Assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Yunli Xing, Dr., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Saczynski JS, McManus DD, Waring ME, Lessard D, Anatchkova MD, Gurwitz JH, Allison J, Ash AS, McManus RH, Parish DC, Goldberg RJ, Kiefe CI. Change in Cognitive Function in the Month After Hospitalization for Acute Coronary Syndromes: Findings From TRACE-CORE (Transition, Risks, and Actions in Coronary Events-Center for Outcomes Research and Education). Circ Cardiovasc Qual Outcomes. 2017 Dec;10(12):e001669. doi: 10.1161/CIRCOUTCOMES.115.001669. PMID 29237744
- [Background] Iadecola C, Yaffe K, Biller J, Bratzke LC, Faraci FM, Gorelick PB, Gulati M, Kamel H, Knopman DS, Launer LJ, Saczynski JS, Seshadri S, Zeki Al Hazzouri A; American Heart Association Council on Hypertension; Council on Clinical Cardiology; Council on Cardiovascular Disease in the Young; Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; and Stroke Council. Impact of Hypertension on Cognitive Function: A Scientific Statement From the American Heart Association. Hypertension. 2016 Dec;68(6):e67-e94. doi: 10.1161/HYP.0000000000000053. Epub 2016 Oct 10. PMID 27977393
- [Background] Sundboll J, Horvath-Puho E, Adelborg K, Schmidt M, Pedersen L, Botker HE, Henderson VW, Sorensen HT. Higher Risk of Vascular Dementia in Myocardial Infarction Survivors. Circulation. 2018 Feb 6;137(6):567-577. doi: 10.1161/CIRCULATIONAHA.117.029127. Epub 2017 Oct 12. PMID 29025764
- [Background] Gu SZ, Beska B, Chan D, Neely D, Batty JA, Adams-Hall J, Mossop H, Qiu W, Kunadian V. Cognitive Decline in Older Patients With Non- ST Elevation Acute Coronary Syndrome. J Am Heart Assoc. 2019 Feb 19;8(4):e011218. doi: 10.1161/JAHA.118.011218. PMID 30773118